CLINICAL TRIAL: NCT00777439
Title: An Investigational New Drug Program for the Use of Domperidone in the Treatment of Refractory Gastroesophageal Reflux Disease and Other Gastrointestinal Motility Disorders
Brief Title: Domperidone for Refractory Gastrointestinal Disorders
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Arnold, George, M.D. (Individual)
Responsible Party: Principal Investigator, George Arnold, MD, Principal Investigator, Arnold, George, M.D.
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GLA102024
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Last update posted 2016-08-18 (Estimated); Status verified 2016-08

CONDITIONS: Gastroparesis
Keywords: Dopamine; Domperidone; Gastroparesis; Gastrointestinal Diseases; Neurologic Manifestations; Stomach Diseases; Digestive System Diseases; Esophagitis; Esophageal Disorders; Paralysis
MeSH Terms: conditions — Gastroparesis; Gastrointestinal Diseases; Neurologic Manifestations; Stomach Diseases; Digestive System Diseases; Esophagitis; Esophageal Diseases; Paralysis | interventions — Domperidone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Domperidone (Other): All eligible subjects will receive domperidone in an open label, single group assignment.
  Interventions: Drug: Domperidone

INTERVENTIONS:
Drug: Domperidone — 10 mg of oral domperidone will be administered 4 times daily. This dose may be increased to 20 mg 4 times daily or 30 mg 4 times daily, depending on how the subject responds to the drug.
  Other Names: Domperidone maleate, Motilium

SUMMARY:
The purpose of this study is to prescribe oral domperidone for subjects with gastrointestinal disorders who have failed or suffered adverse effects from standard medical treatment.

DETAILED DESCRIPTION:
Domperidone is a dopamine-2 receptor antagonist. It acts as a prokinetic agent through its effects on the chemoreceptor trigger zone and the motor function of the stomach and small intestines. It does not cause any adverse neurological symptoms and has an excellent safety profile for long-term oral administration in recommended doses.

In the United States, domperidone is not approved by the Food and Drug Administration (FDA) and cannot be obtained by routine prescriptions or covered by health care insurance plans. It is also illegal to write a prescription for the subject to obtain the drug outside the U.S. Domperidone can be administered legally by obtaining a FDA Investigational New Drug (IND) application with Institutional Review Board (IRB) approval.

This study will follow FDA and IRB regulations and provide domperidone to subjects with gastrointestinal disorders who have failed from standard therapy.

ELIGIBILITY:
Inclusion Criteria:

* Male or female
* Age 18 or older
* Symptoms or manifestations secondary to GERD (e.g., persistent esophagitis, heartburn, upper airway signs or symptoms or respiratory symptoms), gastrointestinal motility disorders such as nausea, vomiting, severe dyspepsia or severe chronic constipation that are refractory to standard therapy.
* Subjects must have a comprehensive evaluation to eliminate other causes of their symptoms.
* Subject has signed informed consent for the administration of domperidone. The informed consent informs the subject of potential adverse events including:

  * increased prolactin levels
  * extrapyramidal side effects
  * breast changes
  * cardiac arrhythmias including QT prolongation
  * there is a potential for increased risk of adverse events with the drugs listed in the addendum

Exclusion Criteria:

* History of or current cardiac disease, including ischemic or valvular heart disease, other structural heart defects, cardiomyopathy or congestive heart failure.
* History of or current arrhythmias including ventricular tachycardia, ventricular fibrillation and Torsade des Pointes. Subjects with minor forms of ectopy (PACs) are not necessarily excluded.
* Clinically significant bradycardia, sinus node dysfunction, or heart block. Prolonged QT syndrome (QTc greater than 450 milliseconds for males, greater 470 milliseconds for females) or family history prolonged QT syndrome.
* Presence of a prolactinoma (prolactin-releasing pituitary tumor).
* Conditions that result in electrolyte disorders, such as severe dehydration, vomiting, malnutrition, eating disorders, renal diseases, or the use of potassium-wasting diuretics or insulin in acute settings. (Note that the presence of vomiting, that may accompany gastroparesis or pseudo- obstruction does not by itself exclude the subject - only if accompanied by electrolyte disturbance must the subject be excluded.)
* Pregnant or breast feeding female.
* Known allergy to domperidone or any components of the domperidone formulation.
* Significantly significant electrolyte disorders.
* Gastrointestinal hemorrhage or obstruction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2008-10; Primary Completion 2017-01 (Estimated); Study Completion 2018-01 (Estimated)

PRIMARY OUTCOMES:
Improvement of symptoms for patients with gastrointestinal disorders who have failed or suffered adverse effects from standard medical treatment. | Domperidone will be prescrided as long as patients benefit from taking it.

CONTACTS AND LOCATIONS:
Overall Officials: George L. Arnold, MD, Principal Investigator — George L. Arnold, MD, FACP
Locations (1):
- Division of Gastroenterology, Hepatology and Nutrition, UPMC Presbyterian Digesive Disorders Center, 3rd Floor, 200 Lothrop Street, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Result] Abell TL, Bernstein RK, Cutts T, Farrugia G, Forster J, Hasler WL, McCallum RW, Olden KW, Parkman HP, Parrish CR, Pasricha PJ, Prather CM, Soffer EE, Twillman R, Vinik AI. Treatment of gastroparesis: a multidisciplinary clinical review. Neurogastroenterol Motil. 2006 Apr;18(4):263-83. doi: 10.1111/j.1365-2982.2006.00760.x. PMID 16553582
- [Result] Barone JA. Domperidone: a peripherally acting dopamine2-receptor antagonist. Ann Pharmacother. 1999 Apr;33(4):429-40. doi: 10.1345/aph.18003. PMID 10332535
- [Result] Ahmad N, Keith-Ferris J, Gooden E, Abell T. Making a case for domperidone in the treatment of gastrointestinal motility disorders. Curr Opin Pharmacol. 2006 Dec;6(6):571-6. doi: 10.1016/j.coph.2006.07.004. Epub 2006 Sep 25. PMID 16997628
- [Result] Reddymasu SC, Soykan I, McCallum RW. Domperidone: review of pharmacology and clinical applications in gastroenterology. Am J Gastroenterol. 2007 Sep;102(9):2036-45. doi: 10.1111/j.1572-0241.2007.01255.x. Epub 2007 May 3. PMID 17488253
- [Result] Soykan I, Sarosiek I, McCallum RW. The effect of chronic oral domperidone therapy on gastrointestinal symptoms, gastric emptying, and quality of life in patients with gastroparesis. Am J Gastroenterol. 1997 Jun;92(6):976-80. PMID 9177513